CLINICAL TRIAL: NCT00094198
Title: Pharmacogenetics and Cardiovascular Events
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1278
Record Dates: First submitted 2004-10-15; First posted 2004-10-15 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Cardiovascular Diseases; Atrial Fibrillation; Cerebrovascular Accident; Heart Diseases; Myocardial Infarction
MeSH Terms: conditions — Cardiovascular Diseases; Atrial Fibrillation; Stroke; Heart Diseases; Myocardial Infarction

SUMMARY:
To assess interactions between selected cardiovascular medications and genes in the incidence of heart attack, stroke, and atrial fibrillation, an irregular heartbeat.

DETAILED DESCRIPTION:
BACKGROUND:

This complex study will collect additional genetic data for 3 ongoing case-control observational studies of drug-gene interactions in myocardial infarction, stroke, and new-onset atrial fibrillation. This study will add single nucleotide polymorphism (SNP) discovery for 16 of 36 candidate genes involving the renin-angiotensin system, sodium transport, adrenergic receptors, and G-proteins, and allow analysis of haplotype data.

The study was initiated in response to RFA HL-03-001, Ancillary Studies in Pharmacogenetics.

DESIGN NARRATIVE:

The primary aim of this study is to assess interactions between selected cardiovascular medications and the major candidate-gene variants or haplotypes on the incidence of myocardial infarction (MI), stroke and atrial fibrillation (AF). The candidate-gene sets-selected on the basis of biology, pharmacology, and information from genome-wide scans-include: (1) 10 genes in the renin-angiotensin system; (2) 10 genes involved in renal sodium transport; (3) 8 genes encoding alpha and beta adrenergic receptors; (4) 8 other genes, including G-proteins, estrogen receptors, and the alpha-1C subunit of the L-type calcium channel. The products of these genes represent the sites of action for many cardiovascular drugs: angiotensin-converting enzyme inhibitors, angiotensin receptor blockers, all classes of diuretics, alpha blockers, beta-blockers, central alpha agonists, calcium antagonists, and estrogens. Both hypothesis-testing and hypothesis-generating analyses are planned. For selected single nucleotide polymorphisms (SNPs) studied in vitro or in small clinical populations, several specific drug-gene interactions are plausible, and these associations will be evaluated in an hypothesis-testing manner.

The study used data from previously funded case-control studies which are expected to produce 1053 MI cases, 565 stroke cases and 800 atrial fibrillation cases and 3249 matching controls from the enrollees of Group Health Cooperative. These patients will already have had chart abstractions, pharmacy database searches, telephone interviews and phlebotomy with specimen storage.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Psaty — University of Washington

REFERENCES:
- [Background] Kooperberg C, Ruczinski I. Identifying interacting SNPs using Monte Carlo logic regression. Genet Epidemiol. 2005 Feb;28(2):157-70. doi: 10.1002/gepi.20042. PMID 15532037
- [Background] Smith NL, Heckbert SR, Lemaitre RN, Reiner AP, Lumley T, Weiss NS, Larson EB, Rosendaal FR, Psaty BM. Esterified estrogens and conjugated equine estrogens and the risk of venous thrombosis. JAMA. 2004 Oct 6;292(13):1581-7. doi: 10.1001/jama.292.13.1581. PMID 15467060
- [Background] Psaty BM, Furberg CD. Contemplating ACTION--long-acting nifedipine in stable angina. Lancet. 2004 Sep 4-10;364(9437):817-8. doi: 10.1016/S0140-6736(04)16992-4. No abstract available. PMID 15351169